CLINICAL TRIAL: NCT06108869
Title: Improving Health and Wellbeing for People Diagnosed With Chronic Spontaneous Urticaria (CSU)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been suspended, as we realised the university still had to finish a contract to provide insurance for myself. Therefore, the recruitment was stopped until this is secured.
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-151
Record Dates: First submitted 2023-10-16; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Intervention Model Description: Single groups will be taken through the ABT programme, or the delayed control intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- 1 (Experimental): 6 Week ABT intervention as described.
  Interventions: Other: ABT Online Programme
- 2 (Experimental): 6 Week ABT intervention as described.
  Interventions: Other: ABT Online Programme
- 3 (Experimental): 6 Week ABT intervention as described.
  Interventions: Other: ABT Online Programme
- 4 (Experimental): 6 Week ABT intervention as described.
  Interventions: Other: ABT Online Programme
- 5 (Experimental): 6 Week ABT intervention as described.
  Interventions: Other: ABT Online Programme
- 6 (Active Comparator): Delayed intervention group
  Interventions: Other: Delayed Control group
- 7 (Active Comparator): Delayed intervention group
  Interventions: Other: Delayed Control group
- 8 (Active Comparator): Delayed intervention group
  Interventions: Other: Delayed Control group
- 9 (Active Comparator): Delayed intervention group
  Interventions: Other: Delayed Control group
- 10 (Active Comparator): Delayed intervention group
  Interventions: Other: Delayed Control group
- 11 (Experimental): ABT intervention as described
  Interventions: Other: ABT Online Programme
- 12 (Experimental): ABT intervention as described
  Interventions: Other: ABT Online Programme
- 13 (Experimental): ABT intervention as described
  Interventions: Other: ABT Online Programme
- 14 (Experimental): ABT intervention as described
  Interventions: Other: ABT Online Programme
- 15 (Experimental): ABT intervention as described
  Interventions: Other: ABT Online Programme
- 16 (Active Comparator): Delayed Control group
  Interventions: Other: Delayed Control group
- 17 (Active Comparator): Delayed Control group
  Interventions: Other: Delayed Control group
- 18 (Active Comparator): Delayed Control group
  Interventions: Other: Delayed Control group
- 19 (Active Comparator): Delayed Control group
  Interventions: Other: Delayed Control group
- 20 (Active Comparator): Delayed Control group
  Interventions: Other: Delayed Control group

INTERVENTIONS:
Other: ABT Online Programme — When the study begins, participants meet each week on Microsoft teams for a 6 week period. Each session will last approximately 1 hour. There will be a maximum of six other participants and two facilitators present at each session. Each session will consist of:
  * A short ABT practice
  * An educational component related to the development of our ABT practice
  * A group discussion on the week's topic and how it relates to you and your diagnosis
  Arms: 1; 11; 12; 13; 14; 15; 2; 3; 4; 5
Other: Delayed Control group — Participants will still meet as a group for first two weeks, before beginning with the ABT practice.
  Arms: 10; 16; 17; 18; 19; 20; 6; 7; 8; 9

SUMMARY:
This study aims to investigate the influence of psychosocial factors on Chronic Spontaneous Urticaria (CSU). Preliminary research suggests a potential link between stress and the experience of CSU symptoms. In light of these findings, our study offers a stress management intervention for individuals diagnosed with CSU.

The intervention consists of a 6-week online course designed to cultivate effective stress management techniques, referred to as 'attention-based training (ABT).' The course asks each participant to develop their own ABT practice, along with a one-hour session per week, providing techniques that participants can use to combat stressors related to their condition.

DETAILED DESCRIPTION:
Chronic Spontaneous Urticaria (CSU) is a common disorder that is poorly understood and frequently misdiagnosed. The burden of the disease can include stress, anxiety, sleep disturbances, and difficulty with activities of daily living. Furthermore, psychological difficulties such as stress, may also aggravate the symptomatic burden of CSU. Holistic interventions are used as a complementary approach to alleviate symptoms in chronic diseases and may represent a valuable non-pharmacological approach in CSU. In 2021, Dr Padraic Dunne and colleagues published a feasibility assessment of an 8 week attention-based training programme to aid in the management of CSU [1]. Whilst this trial was deemed feasible and valuable for participants involved, further research was required with a wider sample to determine the role ABT may have in the management of the condition.

List of Aims and Objectives This current research aims to expand on their pilot study, and provide an evidence based non-pharmacological intervention to aid those in their management of CSU. This project will be the one of the first to provide CSU patients with a psychological intervention in conjunction with their clinical treatment. We believe that a combination of non-pharmacological and pharmacological solutions will ease the suffering caused by this condition and reduce the physical and fiscal burden on the Irish Health service and related clinics.

This study will 1.) Aim to identify the current psychosocial baseline of CSU patients attending urticarial clinics in Ireland and Scotland, to further highlight the psychosocial experience of this population. 2.) Provide and assess the effectiveness of an 6 week ABT programme for CSU management and patient wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Must have diagnosis of CSU

Exclusion Criteria:

* Classified as a vulnerable adult Cannot communicate online, in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Identify Psychosocial Baseline of CSU patents attending Urticaria clinics | 21 months from month 8
  Identify the incidence of abnormal stress/wellbeing scores of CSU patients attending urticarial clinics in Ireland and Scotland, using a baseline questionnaire made up of the Short Stress Overload Scale (10 questions), Five Facet Mindfulness Questionnaire (FFMQ) (39 questions), PERMA Profiler for wellbeing (23 questions), The Urticaria Control Test (4 questions) and Dermatology Life Quality Index (10 questions).
Assess change in psychosocial measures of participants after completing an online 6 week ABT programme | 21 months from month 8
  A psychosocial questionnaire made up of the Short Stress Overload Scale (10 questions), Five Facet Mindfulness Questionnaire (FFMQ) (39 questions), PERMA Profiler for wellbeing (23 questions), The Urticaria Control Test (4 questions) and Dermatology Life Quality Index (10 questions) will be provided to patients pre and post participation in the 6 week online ABT intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Niall Conlon, PhD, Principal Investigator — St. James's Hospital, Ireland
Locations (1):
- St James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 1. Feasibility assessment of an 8-week attention-based training programme in the management of chronic spontaneous urticaria — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-021-00841-z